CLINICAL TRIAL: NCT01844245
Title: Endoscopic Radiofrequency Ablation for Malignant Biliary Strictures Due to Unresectable Cholangiocarcinoma or Ampullary Carcinoma: a Randomised, Controlled, Multicentre Clinical Trial
Brief Title: Endobiliary RFA for Unresectable Malignant Biliary Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bing Hu (Other)
Responsible Party: Sponsor-Investigator, Bing Hu, Professor, Head of Endoscopy Center, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH B-RFA 2013-001
Record Dates: First submitted 2013-04-28; First posted 2013-05-01 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cholangiocarcinoma; Ampullary Carcinoma
Keywords: Cholangiocarcinoma; Ampullary carcinoma; Endoscopic retrograde cholangiopancreatography; Radiofrequency ablation
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endobiliary RFA group (Experimental): 1. Endoscopic retrograde cholangiopancreatography (ERCP) would be performed under standard operating conditions to confirm the biliary malignancy. Subjects will receive endobiliary radiofrequency ablation (Endobiliary RFA) followed by plastic stent(s) placement.
  2. Three months later, subjects will receive the second RFA therapy followed by biliary stents (plastic or SEMS) placement.
  3. During follow-up, if stent occlusion occurs, the patient will undergo endoscopic re-intervention for stent exchange without endobiliary RFA
  Interventions: Procedure: Radiofrequency ablation (RFA)
- Control group (No Intervention): 1. Endoscopic retrograde cholangiopancreatography (ERCP) would be performed under standard operating conditions to confirm the biliary malignancy. Subjects will receive plastic biliary stent(s) placement only.
  2. Three months later, subjects will receive the second endoscopic intervention for stents (plastic or SEMS) exchange.
  3. During follow-up, if stent occlusion occurs, the patient will undergo endoscopic re-intervention for stent exchange without endobiliary RFA

INTERVENTIONS:
Procedure: Radiofrequency ablation (RFA) — The RFA probe is introduced into bile duct. Bipolar electronic coagulation is performed to the tumorous segment.
  Other Names: Endobiliary RFA
  Arms: Endobiliary RFA group

SUMMARY:
Only a small proportion of patients with cholangiocarcinoma or ampullary carcinoma are suitable for surgical resection. The endoscopic or percutaneous transhepatic biliary drainage is accepted approaches for the relief of jaundice in malignant biliary obstruction. But restoration of bile flow have few improvement of the survival of cancer patient. By using endobiliary radiofrequency energy to destruct the tumorous tissue may delay tumour growth, which might improve the survival of patients. The feasibility and safety of this technique using HabibTM EndoHBP probe has been evident. The aims of this randomised, controlled, multicentre study is to evaluate whether endobiliary radiofrequency ablation(RFA) can improve the median survival of patients with unresectable biliary malignancy.

DETAILED DESCRIPTION:
RFA is well established method for treatment of some solid tumors, like liver cancer, lung cancer, etc. Recently, an endoscopically applicable radiofrequency probe, HabibTM EndoHBP catheter, was approved for clinical use. It uses bipolar electrical energy for tissue coagulation and can be easily applied during endoscopic retrograde cholangiopancreatography (ERCP). Endobiliary radiofrequency can destruct the tumor tissue and has potential benefit for controlling tumour growth. Several cohort studies have been published and the feasibility and safety of such technique has been proved.

The aims of this study is to conduct a randomised, controlled, multicentre clinical trial to compare the effect of endobiliary RFA plus biliary stenting with only biliary stenting in patients with unresectable cholangiocarcinoma or ampullary carcinoma.

The objectives are

* To evaluate whether endobiliary RFA prior to biliary stenting can improve the patients' survival as compared to the only stenting therapy.
* To assess the impact of RFA on the stent's patency.

ELIGIBILITY:
Inclusion Criteria:

* Either gender greater than or equal to 18 years of age.
* Cholangiocarcinoma or ampullary cancer unsuitable for surgical resection by staging, comorbidities or patient wishes. Criteria of unresectability being based on 1) metastatic disease or 2) locally advanced.
* Biliary obstruction, Bilirubin > 40umol/L at diagnosis
* Subjects capable of giving informed consent
* Life expectancy of at least 3 months
* Histologically (preferred) or radiologically confirmed cholangiocarcinoma or ampullary cancer

Exclusion Criteria:

* Cardiac Pacemaker
* Patient unstable for endoscopy
* Inability to give informed consent
* Coagulopathy (INR > 2.0 or PTT > 100 sec or platelet count < 50,000)
* Performance status ECOG ≥3 (confined to bed / chair > 50% waking hours)
* Active suppurative cholangitis
* Complex stenoses will not be eligible for the trial
* Patients without access to duodenum or ampulla are not candidates for ERCP and stenting
* Malignant ascites
* Presence of main portal vein thrombosis
* Prior stents placement
* Prior Billroth II or roux-en Y reconstruction
* Inability to insert a guide wire across the malignant stricture
* Pregnancy
* Presence of other malignancy
* Life expectancy < 3months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Patency of stents | 6 months
Unscheduled readmission rates | 6 months
Serious adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bing Hu, MD, PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, The Second Military Medical University
Locations (6):
- China (6):
  - Beijing Friendship Hospital Affiliated to Capital University of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital of the Forth Military Medical University, Xi’an, Shanxi
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Gao DJ, Yang JF, Ma SR, Wu J, Wang TT, Jin HB, Xia MX, Zhang YC, Shen HZ, Ye X, Zhang XF, Hu B. Endoscopic radiofrequency ablation plus plastic stent placement versus stent placement alone for unresectable extrahepatic biliary cancer: a multicenter randomized controlled trial. Gastrointest Endosc. 2021 Jul;94(1):91-100.e2. doi: 10.1016/j.gie.2020.12.016. Epub 2020 Dec 24. PMID 33359435